CLINICAL TRIAL: NCT00450216
Title: A Randomized, Double-Blind, Phase 3 Study of the Efficacy and Safety of HZT-501 in Subjects Requiring NSAID Treatment
Brief Title: Efficacy and Safety Study of HZT-501 in Subjects Requiring Nonsteroidal Anti-Inflammatory Drug (NSAID) Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HZ-CA-303
Record Dates: First submitted 2007-03-19; First posted 2007-03-22 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Ulcer
Keywords: ibuprofen; famotidine; ulcers; NSAIDS; pain; arthritis; chronic regional pain syndrome; chronic soft tissue pain; osteoarthritis; rheumatoid arthritis; chronic low back pain
MeSH Terms: conditions — Ulcer; Pain; Arthritis; Complex Regional Pain Syndromes; Osteoarthritis; Arthritis, Rheumatoid | interventions — Ibuprofen; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): HZT-501: Ibuprofen 800mg/famotidine 26.6mg
  Interventions: Drug: Ibuprofen/famotidine
- 2 (Active Comparator): Ibuprofen 800mg
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen/famotidine — HZT-501: Ibuprofen800mg/famotidine 26.6mg administered orally 3 times daily for 24 weeks
  Arms: 1
Drug: Ibuprofen — Ibuprofen 800mg administered orally 3 times daily for 24 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate whether HZT-501 is effective in reducing the rate of development of ibuprofen-associated ulcers in patients who require long-term daily use of ibuprofen.

DETAILED DESCRIPTION:
HZT-501 is a combination product including ibuprofen and the acid reducing agent famotidine. The study is designed to determine whether the combination product reduces the rate of ulcer development in subjects who require long-term daily use of ibuprofen.

Subjects will be assigned randomly, in approximately a 2:1 ratio, to treatment with either HZT-501 (ibuprofen 800 mg/famotidine 26.6 mg) or ibuprofen (800 mg) three times daily for a 24 week treatment period or until they develop either an endoscopically-diagnosed upper gastrointestinal ulcer and/or prohibitive toxicity. Subjects will visit the study center for Screening and at Weeks 4, 8, 16, and 24. Physical exams will be performed, and clinical laboratory measurements made, at selected times during the study. Endoscopic exams will be performed during Screening and at Weeks 8, 16, and 24. Subjects will be contacted four weeks following study completion.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Expected to require daily administration of an NSAID for at least the coming six months for conditions such as osteoarthritis, rheumatoid arthritis, chronic low back pain, chronic regional pain syndrome, and chronic soft tissue pain.
* Did not use a NSAID within the 30 days prior to study entry

Exclusion Criteria:

* History of erosive esophagitis
* History of any of the following serious gastrointestinal complications:

  * perforation of ulcers,
  * gastric outlet obstruction due to ulcers, or
  * gastrointestinal bleeding.
* Active cardiac, renal, and/or hepatic disease
* Current Helicobacter pylori (H. pylori) infection
* Use of an acid suppressant agent, misoprostol, or more than 325 mg/day of aspirin within the 14 days prior to study entry.
* Uncontrolled diabetes
* Uncontrolled hypertension
* Positive pregnancy test at screening
* Positive test at Screening for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* Currently participating, or participation within 30 days prior to study entry, in an investigational drug study

Please note that there are other additional criteria. The study center will determine if patients meet all of the criteria.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 906 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Bello AE, Kent JD, Holt RJ. Gastroprotective efficacy and safety of single-tablet ibuprofen/famotidine vs ibuprofen in older persons. Phys Sportsmed. 2015 Jul;43(3):193-9. doi: 10.1080/00913847.2015.1066229. Epub 2015 Jul 13. PMID 26165391

RESULTS

PARTICIPANT FLOW:
Groups:
- HZT-501: HZT-501: Ibuprofen 800mg/famotidine 26.6mg tablets t.i.d.
- Ibuprofen: Ibuprofen 800mg tablets t.i.d.
Period: Overall Study
Arm/Group | HZT-501 | Ibuprofen
Started | 607 | 299
Completed | 433 | 170
Not Completed | 174 | 129
Not completed — Adverse Event | 38 | 23
Not completed — Withdrawal by Subject | 48 | 26
Not completed — Lost to Follow-up | 16 | 9
Not completed — upper gastrointestinal (UGI) ulcer | 51 | 51
Not completed — misc | 21 | 20

BASELINE CHARACTERISTICS:
Groups:
- HZT-501: HZT-501: Ibuprofen 800mg/famotidine 26.6mg
- Ibuprofen: Ibuprofen 800mg
- Total: Total of all reporting groups
Arm/Group | HZT-501 | Ibuprofen | Total
Number analyzed (Participants) | 607 | 299 | 906
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 500 | 240 | 740
  >=65 years | 107 | 59 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (9.2) | 55.9 (9.3) | 55.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 416 | 208 | 624
  Male | 191 | 91 | 282
Region of Enrollment [Number; unit: participants]
  United States | 607 | 299 | 906

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Develop Endoscopically-diagnosed Gastric Ulcers
Description: The primary efficacy endpoint was the number of participants with gastric ulcer at any time throughout 24 weeks of treatment. An ulcer was defined as a mucosal break of at least 3 mm in diameter with unequivocal depth. A participant is considered to have completed the study if all scheduled assessments up through the Week 24 visit have been performed.
Time Frame: 24 weeks
Population: All randomized participants who received at least one dose of study drug and who underwent a baseline endoscopic examination and at least the Week 8 endoscopic examination. Participants were assigned according to the treatment to which they were randomized; 2:1 randomization, HZT-501:ibuprofen.
Measure: Number; unit: participants
Arm/Group | HZT-501 | Ibuprofen
Number analyzed (Participants) | 550 | 262
participants | 55 [4.4 to 15.3] | 52 [4.4 to 15.3]
Statistical Analysis 1: Comparison: HZT-501 vs Ibuprofen; The primary efficacy endpoint was the number of participants developing gastric ulcers throughout 24 weeks of treatment. A summary, including cumulative frequency and percentage with associated 95% confidence intervals was produced for the observational incidences of gastric ulcers at 24 weeks. The cumulative number of participants developing gastric ulcers at 24 weeks was analyzed using the Cochran-Mantel-Haenszel (CMH) test stratified by use of low-dose aspirin and prior UGI ulcer history; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — CMH test stratified by use of low-dose aspirin (yes/no) and prior upper gastrointestinal (UGI) ulcer history (yes/no) at randomization; Risk Difference (RD) = 9.8, 95% CI 2-sided [4.4 to 15.3]

2. Secondary Outcome: Number of Participants Who Develop Endoscopically-diagnosed Upper Gastrointestinal (UGI) Ulcers During the 24-week Treatment Period.
Description: The secondary efficacy endpoint was the number of participants with UGI (i.e., gastric and/or duodenal) ulcer at any time throughout 24 weeks of treatment. An ulcer was defined as a mucosal break of at least 3 mm in diameter with unequivocal depth. A participant is considered to have completed the study if all scheduled assessments up through the Week 24 visit have been performed.
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | HZT-501 | Ibuprofen
Number analyzed (Participants) | 550 | 262
participants | 63 [6.1 to 17.6] | 61 [6.1 to 17.6]
Statistical Analysis 1: Comparison: HZT-501 vs Ibuprofen; The secondary efficacy endpoint was the number of participants developing UGI (i.e., gastric and/or duodenal) ulcers throughout 24 weeks of treatment. A summary, including cumulative frequency and percentage with associated 95% confidence intervals was produced for the observational incidences of UGI ulcers at 24 weeks. The cumulative number of participants developing UGI ulcers at 24 weeks was analyzed using the CMH test stratified by use of low-dose aspirin and prior UGI ulcer history; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — CMH test stratified by use of low-dose aspirin (yes/no) and prior UGI ulcer history (yes/no) at randomization; Risk Difference (RD) = 11.8, 95% CI 2-sided [6.1 to 17.6]

3. Secondary Outcome: Number of Participants Who Develop Endoscopically-diagnosed Duodenal Ulcers During the 24-week Treatment Period.
Description: The secondary efficacy endpoint was the number of participants with duodenal ulcer at any time throughout 24 weeks of treatment. An ulcer was defined as a mucosal break of at least 3 mm in diameter with unequivocal depth. A participant is considered to have completed the study if all scheduled assessments up through the Week 24 visit have been performed.
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | HZT-501 | Ibuprofen
Number analyzed (Participants) | 550 | 262
participants | 8 [1.0 to 6.8] | 14 [1.0 to 6.8]
Statistical Analysis 1: Comparison: HZT-501 vs Ibuprofen; The secondary efficacy endpoint was the number of participants developing duodenal ulcers throughout 24 weeks of treatment. A summary, including cumulative frequency and percentage with associated 95% confidence intervals was produced for the observational incidences of duodenal ulcers at 24 weeks. The cumulative number of participants developing duodenal ulcers at 24 weeks was analyzed using the CMH test stratified by use of low-dose aspirin and prio UGI ulcer history at randomization; Test type: Superiority or Other; p = 0.0006, Cochran-Mantel-Haenszel — CMH test stratified by use of low-dose aspirin (yes/no) and prior UGI ulcer history (yes/no) at randomization; Risk Difference (RD) = 3.8, 95% CI 2-sided [1.0 to 6.8]

4. Secondary Outcome: The Number of Participants Developing Non-steroidal Anti-inflammatory (NSAID)Associated Serious Gastrointestinal Complications (Perforation of Ulcers, Gastric Outlet Obstruction Due to Ulcers, Gastrointestinal Bleeding)
Description: The secondary efficacy endpoint was the number of participants developing a NSAID-associated serious gastrointestinal complication at any time throughout 24 weeks of treatment. A NSAID-associated serious gastrointestinal complication was defined as a perforation of ulcers, gastric outlet obstruction due to ulcers, and/or gastrointestinal bleeding.
Time Frame: 24 weeks
Measure: Number; unit: particpants
Arm/Group | HZT-501 | Ibuprofen
Number analyzed (Participants) | 550 | 262
particpants | 3 | 0

ADVERSE EVENTS:
Time Frame: Randomization to 28 weeks.
Description: Safety Population: All randomized participants who received at least one dose of study drug and who underwent a baseline endoscopic examination. Participants were assigned to the treatment to which they received; 2:1 randomization, HZT-501:ibuprofen.
Arm/Group | HZT-501 | Ibuprofen
Serious Adverse Events (participants affected / at risk) | 22/607 | 13/299
Other Adverse Events (participants affected / at risk) | 342/607 | 184/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HZT-501 (N=607) | Ibuprofen (N=299)
abdominal hernia (Gastrointestinal disorders) | 1 | 0
alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
bipolar disorder (Psychiatric disorders) | 0 | 1
blood creatinine increased (Investigations) | 1 | 0
bronchits (Infections and infestations) | 0 | 1
calculus ureteric (Renal and urinary disorders) | 1 | 0
cardio-respiratory arrest (Cardiac disorders) | 0 | 2
cellulits (Infections and infestations) | 2 | 0
chest pain (General disorders) | 2 | 1
cholecystitis (Hepatobiliary disorders) | 1 | 0
coronary artery disease (Cardiac disorders) | 0 | 1
dehydration (Metabolism and nutrition disorders) | 2 | 0
depression (Psychiatric disorders) | 1 | 1
drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
esoinophilia (Blood and lymphatic system disorders) | 0 | 1
hemorrhoid hemorrhage (Gastrointestinal disorders) | 1 | 0
hemorrhoids (Gastrointestinal disorders) | 1 | 0
hypertension (Vascular disorders) | 1 | 0
hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
major depression (Psychiatric disorders) | 1 | 0
menorrhagia (Reproductive system and breast disorders) | 1 | 0
migraine (Nervous system disorders) | 1 | 0
multi-organ failure (General disorders) | 0 | 1
myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
non-cardiac chest pain (General disorders) | 1 | 0
osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
pneumonia (Infections and infestations) | 1 | 2
renal failure acute (Renal and urinary disorders) | 3 | 0
road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
schizoaffective disorder (Psychiatric disorders) | 1 | 0
syncope (Nervous system disorders) | 0 | 1
traumatic brain injury (Injury, poisoning and procedural complications) | 2 | 1
upper respiratory tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HZT-501 (N=607) | Ibuprofen (N=299)
abdominal distension (Gastrointestinal disorders) | 4 | 5
abdominal pain (Gastrointestinal disorders) | 8 | 4
abdominal pain upper (Gastrointestinal disorders) | 20 | 7
abdominal tenderness (Gastrointestinal disorders) | 5 | 4
anemia (Blood and lymphatic system disorders) | 13 | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 6
back pain (Musculoskeletal and connective tissue disorders) | 8 | 1
blood pressure increased (Investigations) | 6 | 2
bronchitis (Infections and infestations) | 13 | 4
constipation (Gastrointestinal disorders) | 27 | 13
contusion (Injury, poisoning and procedural complications) | 2 | 4
cough (Respiratory, thoracic and mediastinal disorders) | 12 | 9
diarrhea (Gastrointestinal disorders) | 30 | 13
dizziness (Nervous system disorders) | 9 | 5
dry mouth (Gastrointestinal disorders) | 6 | 2
dyspepsia (Gastrointestinal disorders) | 31 | 23
edema peripheral (General disorders) | 14 | 6
epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 0
fall (Injury, poisoning and procedural complications) | 5 | 4
fatigue (General disorders) | 2 | 4
flatulence (Gastrointestinal disorders) | 8 | 2
gastritis (Gastrointestinal disorders) | 3 | 4
gastroenteritis viral (Infections and infestations) | 8 | 1
gastroesophageal reflux disease (Gastrointestinal disorders) | 10 | 8
headache (Nervous system disorders) | 23 | 9
herpes zoster (Infections and infestations) | 3 | 3
hypertension (Vascular disorders) | 21 | 7
influenza (Infections and infestations) | 9 | 7
insomnia (Psychiatric disorders) | 7 | 1
muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 2
nasopharyngitis (Infections and infestations) | 12 | 8
nausea (Gastrointestinal disorders) | 40 | 13
neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3
pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 3
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 4
pneumonia (Infections and infestations) | 3 | 4
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 4
sinusitis (Infections and infestations) | 12 | 11
stomach discomfort (Gastrointestinal disorders) | 14 | 4
syncope (Nervous system disorders) | 3 | 3
toothache (Gastrointestinal disorders) | 3 | 3
upper respiratory tract infection (Infections and infestations) | 23 | 10
urinary tract infection (Infections and infestations) | 14 | 9
viral upper respiratory tract infection (Infections and infestations) | 3 | 3
vomiting (Gastrointestinal disorders) | 15 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI reserves the right to publish or otherwise make public the Study results provided that such communication occurs only after (i) the results of the multicenter Study in its entirety have been publicly disclosed by, or with consent of the sponsor or (ii) 18 months after conclusion of the Study at all sites, whichever comes first. Following this, PI can publish, present or use any non-confidential study results following Sponsor review. PI will not make public raw data or Case Reports.